CLINICAL TRIAL: NCT06812624
Title: The Effect of Perioperative Results on Mortality in Coronary Artery Bypass Surgery: Risk Assessment with Fuzzy Logic
Brief Title: The Effect of Perioperative Results on Mortality in Coronary Artery Bypass Surgery
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kerem Erkalp, MD, Prof, professor, Istanbul University - Cerrahpasa
Other Study IDs: 112
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases; Cardiovascular Complication; Anesthesia
Keywords: Fuzzy logic; mortality; coronary artery surgery; risk assessment; risk scoring system; complications
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- coronary artery bypass surgery group: All patients over the age of 18 who underwent isolated coronary artery bypass surgery at the IUC Cardiology Institute hospital between January 1, 2020 and July 31, 2024 will be included in the study.
  Interventions: Other: There is no intervention in this study.

INTERVENTIONS:
Other: There is no intervention in this study. — This study is planned as a retrospective cross sectional study. Only the information of the patients will be used.

SUMMARY:
Coronary artery bypass grafting (CABG) is one of the most common heart surgeries. Most patients are elderly with comorbidities that affect morbidity and mortality rates. Even in developed countries mortality rate is 1.9-5.3%. Determination of perioperative risk factors and creating protocols to take precautions accordingly may reduce mortality in patients.

In CABG patients, due to the surgical burden combined with existing comorbidities, it is important for physicians to evaluate the risk status and predict the mortality rates. For this purpose, various scoring systems have been developed.

Fuzzy logic method allows partially membership, so that a glass that is neither full nor empty can be numerically expressed as being partially full but also partially empty. This feature is similar to the reasoning structure of the human brain that uses linguistic tools. In this way, in cases where there is no precise mathematical model and where the existence of imprecise and uncertain information is natural, such as medical applications, in order to solve the problem, fuzzy easily allows linguistic expressions containing the knowledge, experience and intuition of expert to transforme into the model created for the solution. In decision making process, fuzzy logic provides ability to use linguistic expressions, including experts' intuition. Thus, decisions can be made even with approximate data and uncertainty. For this reason, fuzzy logic is used in a wide range of research from engineering to medicine.

The records of patients who underwent CABG surgery in Istanbul University-Cerrahpaşa Cardiology Institute between January 1, 2020 and July 31, 2024 will be examined.

Preoperative major risk factors diabetes, pulmonary, neurological, kidney and liver disease with preoperative minor risk factors age, weight and smoking will be recorded. Perioperative risk factors; duration of artificial circulation, number of vessels bypassed, and number of blood products used will be recorded. Our primary aim is to create a fuzzy logic-based perioperative risk classification model to identify high-risk patients in CABG surgery. Secondly we aimed to investigate the effect of perioperative risk factors on postoperative complications

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) is one of the most common heart surgeries. Most patients are elderly with comorbidities such as diabetes mellitus and renal diseases. Tehese risk factors affect morbidity and mortality rates. Even in developed countries mortality rate in CABG patients is between 1.9-5.3%. Identifying perioperative risk factors and taking precautions by creating protocols can decrease mortality in patients. Experienced surgical and anesthesia teams, evidence-based practices, and advances in pharmacology and technology can increase survival.

Risk assessment is important in determining the treatment plans of patients who will be operated on, providing patient education for the postoperative period, providing insight into prognosis, and determining health care quality standards.

In CABG patients, due to the surgical burden combined with existing comorbidities, it is important for physicians to evaluate the risk status and predict the mortality rates. For this purpose low and high risk studies have been conducted and various scoring systems have been developed. European System for Cardiac Operative Risk Evaluation-II (EUROSCORE-II) is a scoring system that was created specifically for cardiac surgery patients and is widely used all over the world, predicting mortality through preoperative evaluation. EUROSCORE-II scoring may be low in older patients (over 70 years of age). A scoring system with higher predictive power is aimed by making modifications to EUROSCORE-II or comparisons with other scoring systems.

In 1965, Zadeh first introduced Fuzzy, which is the basis of the fuzzy logic procedure Fuzzy logic method allows partially membership, so that a glass that is neither full nor empty can be numerically expressed as being partially full but also partially empty. This feature is similar to the reasoning structure of the human brain that uses linguistic tools. In this way, in cases where there is no precise mathematical model and where the existence of imprecise and uncertain information is natural, such as medical applications, in order to solve the problem, fuzzy easily allows linguistic expressions containing the knowledge, experience and intuition of expert to transforme into the model created for the solution. In decision making process, fuzzy logic provides ability to use linguistic expressions, including experts' intuition. Thus, decisions can be made even with approximate data and uncertainty. For this reason, fuzzy logic is used in a wide range of research from engineering to medicine.

The records of patients who underwent isolated CABG surgery in Istanbul University-Cerrahpaşa Cardiology Institute between January 1, 2020 and July 31, 2024 will be included.

Diabetes mellitus, pulmonary, neurological, kidney and liver disease will be recorded as preoperative major risk factors. Age, weight and smoking will be recorded as preoperative minor risk factors. Duration of artificial circulation, number of vessels bypassed, and number of blood products used will be recorded as perioperative risk factors.

The effect of preoperative risk factors on mortality has been investigated in many studies. Our primary aim is to create a fuzzy logic-based perioperative risk classification model to identify high-risk patients in isolated CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* All isolated coronary artery bypass surgery between January 1, 2020 and July 31, 2024 at IUC Cardiology Institute hospital

Exclusion Criteria:

* All surgical procedures other than isolated coronary artery bypass surgery and patients under the age of 18 were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over 18 year of age, all isolated coronary artery bypass surgery between January 1, 2020 and July 31, 2024 at IUC Cardiology Institute hospital
Sampling Method: Probability Sample
Enrollment: 485 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Risk assessment with fuzzy logic | 4 months
  Create a fuzzy logic-based perioperative risk classification model to identify high-risk patients in CABG operations.

SECONDARY OUTCOMES:
Perioperative risk factors | 4 months
  Investigate the effects of artificial circulation time, number of bypassed vessels, and how many bags of blood products were used as perioperative risk factors on postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Kerem Erkalp, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)